CLINICAL TRIAL: NCT01556503
Title: Sensitivity/Specificity Study of Non-invasive Imaging for Melanoma Diagnosis
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006939; CPC-11033-L (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2012-03-12; First posted 2012-03-16 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pigmented Lesion: Patients identified as having a concerning pigmented lesion and the physician believes it is appropriate to biopsy to rule out melanoma.
  Interventions: Device: VivaScope System

INTERVENTIONS:
Device: VivaScope System — VivaScope System, Model#s 1500 and 2500
  Other Names: Confocal Microscope

SUMMARY:
The purpose of this study is to show how well a new device, confocal microscope, works to detect malignant melanoma, a type of skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 or older
* Patient who has already been selected by their dermatologist for biopsy of a suspicious pigmented lesion and who consents to participate in the study
* Signed informed consent

Exclusion Criteria:

* Age < 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity of confocal microscope to improve melanoma detection | Up to 1 year
  Determine the sensitivity of confocal microscopy in the diagnosis of melanoma by comparison to the gold standard histopathologic diagnosis.
Specificity of the confocal microscope to improve melanoma detection | Up to 1 year
  Determine the specificity of confocal microscopy in the diagnosis of melanoma by comparison to the gold standard histopathologic diagnosis

SECONDARY OUTCOMES:
Patterns seen on the confocal image | Up to 1 year
  Evaluate and confirm patterns seen on the confocal image, which are characteristic of melanoma and atypical nevi:
  A) Pagetoid melanoma cells: melanocytes in suprabasal areas of the epidermis B) Irregular dermal-epidermal junction

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simpson, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States